CLINICAL TRIAL: NCT04964310
Title: Pharmacogenomics of APAP Induced DILI in Chinese Population.
Brief Title: Screening of Susceptibility Genes for APAP Induced Drug Induced LIver Injury in ChiNese Population: a Case-control Study
Acronym: PAIN
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: University of Colorado, Denver (Other); Beijing Genomics Institute (Other); Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Hao Sun, associate professor, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Other Study IDs: FirstNanjingMUED
Record Dates: First submitted 2021-07-07; First posted 2021-07-16 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Acetaminophen; Drug-Induced Liver Injury; Pharmacogenetics; China
Keywords: Acetaminophen; Drug-Induced Liver Injury; Pharmacogenetics; China; Case-Control Studies; candidate gene
MeSH Terms: conditions — Chemical and Drug Induced Liver Injury | interventions — Polymorphism, Genetic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — whole blood for DNA extraction
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- APAP_DILI: （①/②）+③+④：
  ① history of acetaminophen exposure ② abnormal acetaminophen concentration in blood or urine：≥150µg/mL after 4 hour ，≥4.5µg/mL at anytime，measurable ≥24 hours③ liver impairment：Alanine aminotransferase (ALT) or Aspartate Aminotransferase (AST) ≥ 1000 IU/L ④ liver impairment is caused by acetaminophen：Russel U-Calf Causality Assessment Method(RUCAM) causality score>6
  Interventions: Genetic: genetic polymorphism
- APAP_NO-DILI（NDILI）: （①/②）not（③/④）：
  ① history of acetaminophen exposure ② abnormal acetaminophen concentration in blood or urine：≥150µg/mL after 4 hour ，≥4.5µg/mL at anytime，measurable ≥24 hours③ liver impairment：ALT or AST ≥ 1000 IU/L④ liver impairment is caused by acetaminophen：RUCAM causality score>6

INTERVENTIONS:
Genetic: genetic polymorphism — Observe the genetic polymorphism frequency difference between case and control groups
  Groups: APAP_DILI

SUMMARY:
Acetaminophen (APAP) is the most commonly used NSAIDS in clinic, and it is also a common cause of drug-induced liver injury (DILI). In 2012, the proportion of DILI caused by APAP in the United States was 51%, while in Asia, it was only 7.10%. Previously, a small cohort study in the United States screened for some of the susceptibility genes for DILI due to APAP by the Genome wide association study (GWAS) method. However, the genetic susceptibility loci based on the US cohort were not applicable to the Chinese population. Therefore, we make a study design include Chinese population who ingested APAP and divided them into case group and control group according to the occurrence of DILI. We hope to be able to find the root of differences at the genetic level and explore new pathogenic mechanisms.

DETAILED DESCRIPTION:
I. Study Object

(i) Into the group strategy: continuous into group.

(ii) Grouping strategy：

1. Case group.

   Inclusion criteria：
   * A clear history of acetaminophen (or acetaminophen-containing drugs) ingestion.
   * Plasma and/or urine testing for acetaminophen components if history of ingestion is unclear.
   * Monitoring of Alanine aminotransferase (ALT) or Aspartate Aminotransferase (AST) ≥ 1000 IU/L at any time after APAP administration and Roussel Causality Assessment Method(RUCAM) score > 6
   * Age ≥ 14 years old.
   * The subject or guardian agrees to participate in this project and signs an informed consent form.

   Exclusion criteria： •The use of drugs for which frequency of adverse reactions to liver damage is defined as "common or very common" (≥1%) in the instructions.
   * Concurrent use of herbs that are clearly susceptible to liver damage (see list of definitions in the Annex).
   * Have a known definite cause of liver damage: active viral hepatitis; alcoholic liver disease; autoimmune liver disease; primary or secondary liver tumors; and other underlying liver disease that has affected liver function.
   * Those who fail to provide complete general information and clinical information.
   * Subjects or guardians who do not agree to see this project do not sign the informed consent form.
2. Control group

   Inclusion criteria：
   * A clear history of acetaminophen (or acetaminophen-containing drugs) ingestion.
   * Plasma and/or urine testing for acetaminophen components if history of APAP ingestion is unclear.
   * Age: ≥ 14 years old.
   * The subject or guardian agrees to participate in this project and signs an informed consent form.

   Exclusion criteria： •The use of drugs for which frequency of adverse reactions to liver damage is defined as "common or very common" (≥1%) in the instructions.

   •Concurrent use of herbs that are clearly susceptible to liver damage (see list of definitions in the Annex).

   •There are known definite causes of liver damage (see attached list of definitions): active viral hepatitis; alcoholic liver disease; autoimmune liver disease; primary or secondary liver tumors; and other underlying liver disease that has affected liver function.

   •Those who fail to provide complete general information and clinical information.

   •Subjects or guardians who do not agree to see this project do not sign the informed consent form.

   (iii) Matching strategy.

   Matching principle：

   •Case and control participants were matched according to ingested dose, duration of antidote administration, and duration of gastric lavage.

   •1:2 matching.

   Confounding factors：

   •Dose intake: patient report (primary) + blood concentration test (secondary)

   •Antidote use time: <4 hours, 4-24 hours, >24 hours

   •Gastric lavage time: <1 hour, ≥1 hour

   (iv) Estimation of sample size

   Parameter source：
   * Focus on drug metabolizing enzymes, immunogenic loci
   * The distribution of APAP-dependent DILI susceptibility allele frequencies in Asian populations based on literature findings.

2. Parameter value：

* Hypothesis: Gene-Environment.
* Outcome Model: Baseline risk P0=0.10.
* Genetic Effect =1.2,
* Power=0.8, Type I error rate=0.05 (two-sided).

Results： The case sample size should be 113 with a control sample size of 226.

II. Exposure/risk factors.

(i) Definition. Exposure factors refer to susceptibility genes for DILI caused by APAP, including：

* 2,036,060 marker sites
* Human Leukocyte Antigen (HLA) :HLA-A and HLA-B immune loci.
* Genotype-Imputation.

(ii) Measurement methods.

1. Adopt candidate gene strategy. The candidate gene strategy is a flexible approach with low cost, relatively simple quality control and statistical analysis, and a relatively easy biological explanation behind the association because the genes selected are all important for the disease.
2. Using the hypothesis-driven approach. Considering the hypothesis that some specific genes may be associated with the study outcome, a sequence-based approach was chosen for the analysis of potentially functional single nucleotide polymorphism (SNPs), selecting SNPs that are more likely to be of functional value associated with drug metabolizing enzymes, immunogenic loci, drug transport proteins, drug-acting receptors and other links, especially those located in candidate genes coding regions.
3. Using custom chips. The Expanded Multi-Ethnic Genotyping Array (MEGAEX), a microarray built by consortia with enhanced capabilities to understand complex diseases in a variety of populations. This commercially available microarray determines individual drug response through the detection of 2,036,060 marker loci. It also complements HLA-A and HLA-B immune loci information to complete Genotype-Imputation.

III. Quality control The study has a strict standard test operation procedure, and relevant training is conducted for the personnel involved in the test before the start of the experiment, and the test can only be conducted after passing the training. We have a quality control center with dedicated personnel responsible for subject progress and data quality control. An online digital randomization platform and information entry management system is set up based on the web server terminal, which is capable of timely case randomization grouping and electronic clinical case observation form information entry, and can effectively and automatically check and correct errors during the information entry process. That is, it helps to ensure the accuracy and reliability of the entered information, and can provide real-time data monitoring for the supervisors. In addition, this study will monitor the conduct of experiments and data entry.

IV. Data Management Plan

* Data Center: The data management center established by the national data management standard undertakes data management work.
* Data management system: REDCap is used to establish electronic case report forms for online data collection and management.
* Data collection: Data entry by independent data registrants not involved in the study in the study lead unit.
* Data consistency monitoring: Data consistency monitoring by an independent third-party monitor.
* Data audit and locking: Data is audited, cleaned and locked by a dedicated data manager.

V. Statistical analysis plan

(i) Hypothesis testing. H0: No difference in genes between subjects with and without liver damage after ingestion of APAP H1: Significant genetic differences between subjects with and without liver damage after ingestion of APAP

(ii) Analytical strategies.

* Continuous variables were described as mean ± standard deviation (SD) or median of interquartile range (IQR), and differences between groups were analyzed by two-factor ANOVA or nonparametric tests. Categorical variables were expressed as numbers and percentages and analyzed by logistic regression models.
* Hardy-Weinberg equilibrium (HWE) between control groups was tested using the goodness-of-fit χ2 test. Using haplotype analysis view（Haploview） 4.2 software, the haplotype region group was selected considering the linkage disequilibrium between tags of single nucleotide polymorphisms (tagSNPs).
* Multivariate conditional logistic regression analysis was performed to estimate the association between genotype and risk of DILI from APAP by dominance ratios (ORs) and 95% confidence intervals (CIs) with gastric lavage and antidote use as covariates.
* Three different genetic models were used to synthesize the role of tagSNPs. Software package for Hardy-weinberg analysis(SHEsis) online program was used for haplotype analysis under logistic regression model.
* All analyses were performed using Statistics is a powerful statistical software platform(SPSS) for Windows (version 26.0 USA). Two-tailed P values <0.05 were considered statistically significant.

ELIGIBILITY:
Inclusion criteria：

* A clear history of acetaminophen (or acetaminophen-containing drugs) ingestion.
* Plasma and/or urine testing for acetaminophen components if history of ingestion is unclear.
* Monitoring of Alanine aminotransferase (ALT) or Aspartate Aminotransferase (AST) ≥ 1000 IU/L at any time after APAP administration and Roussel Uclaf Causality Assessment Method(RUCAM) score > 6
* Age ≥ 14 years old
* The subject or guardian agrees to participate in this project and signs an informed consent form.

Exclusion criteria：

* The use of drugs for which frequency of adverse reactions to liver damage is defined as "common or very common" (≥1%) in the instructions.
* Concurrent use of herbs that are clearly susceptible to liver damage (see list of definitions in the Annex).
* Have a known definite cause of liver damage: active viral hepatitis; alcoholic liver disease; autoimmune liver disease; primary or secondary liver tumors; and other underlying liver disease that has affected liver function.
* Those who fail to provide complete general information and clinical information.
* Subjects or guardians who do not agree to see this project do not sign the informed consent form.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: history of acetaminophen exposure
Sampling Method: Non-Probability Sample
Enrollment: 339 (Estimated)
Dates: Start 2020-08-31 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
genetic polymorphism | 2 year
  the genetic polymorphism（HLA、SNPs ）frequency difference between case and control groups

CONTACTS AND LOCATIONS:
Overall Officials: Jingsong Zhang, professor, Study Chair — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Danan G, Teschke R. RUCAM in Drug and Herb Induced Liver Injury: The Update. Int J Mol Sci. 2015 Dec 24;17(1):14. doi: 10.3390/ijms17010014. PMID 26712744
- [Background] Major JM, Zhou EH, Wong HL, Trinidad JP, Pham TM, Mehta H, Ding Y, Staffa JA, Iyasu S, Wang C, Willy ME. Trends in rates of acetaminophen-related adverse events in the United States. Pharmacoepidemiol Drug Saf. 2016 May;25(5):590-8. doi: 10.1002/pds.3906. Epub 2015 Nov 3. PMID 26530380
- [Background] Bower WA, Johns M, Margolis HS, Williams IT, Bell BP. Population-based surveillance for acute liver failure. Am J Gastroenterol. 2007 Nov;102(11):2459-63. doi: 10.1111/j.1572-0241.2007.01388.x. Epub 2007 Jun 29. PMID 17608778
- [Background] Chiew AL, Reith D, Pomerleau A, Wong A, Isoardi KZ, Soderstrom J, Buckley NA. Updated guidelines for the management of paracetamol poisoning in Australia and New Zealand. Med J Aust. 2020 Mar;212(4):175-183. doi: 10.5694/mja2.50428. Epub 2019 Dec 1. PMID 31786822
- [Background] Smilkstein MJ, Knapp GL, Kulig KW, Rumack BH. Efficacy of oral N-acetylcysteine in the treatment of acetaminophen overdose. Analysis of the national multicenter study (1976 to 1985). N Engl J Med. 1988 Dec 15;319(24):1557-62. doi: 10.1056/NEJM198812153192401. PMID 3059186
- [Background] Leventhal TM, Gottfried M, Olson JC, Subramanian RM, Hameed B, Lee WM; Acute Liver Failure Study Group. Acetaminophen is Undetectable in Plasma From More Than Half of Patients Believed to Have Acute Liver Failure Due to Overdose. Clin Gastroenterol Hepatol. 2019 Sep;17(10):2110-2116. doi: 10.1016/j.cgh.2019.01.040. Epub 2019 Feb 5. PMID 30731196
- [Background] Lammers LA, Achterbergh R, Pistorius MC, Romijn JA, Mathot RA. Quantitative Method for Simultaneous Analysis of Acetaminophen and 6 Metabolites. Ther Drug Monit. 2017 Apr;39(2):172-179. doi: 10.1097/FTD.0000000000000373. PMID 28045783
- [Background] Monte AA, Sonn B, Saben J, Rumack BH, Reynolds KM, Dart RC, Heard KJ. The Genomics of Elevated ALT and Adducts in Therapeutic Acetaminophen Treatment: a Pilot Study. J Med Toxicol. 2021 Apr;17(2):160-167. doi: 10.1007/s13181-020-00815-2. Epub 2020 Oct 13. PMID 33051802